CLINICAL TRIAL: NCT01278524
Title: International Multicenter Study One Day Prevalence Observational Study for Delirium on ICU
Acronym: IMPROVE-ICU
Status: Completed | Type: Observational
Sponsor: Claudia Spies (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Prof. Dr. C. Spies, MD, Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: IMPROVE-ICU
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Delirium
Keywords: Delirium; Analgosedation; ICU; Pain; Implementation
MeSH Terms: conditions — Delirium; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients: Patients staying in the ICU on the 25th of January

SUMMARY:
An anonymous international multicenter - clinical survey, one-day observational study.

DETAILED DESCRIPTION:
Delirium is a serious complication in postoperative and critically ill patients and is independently associated with cognitive impairment at hospital discharge and with significantly higher 6-month mortality. Furthermore, ICU delirium is associated with more days requiring mechanically ventilation, longer ICU length of stay, and longer hospital length of stay. More recently a study by Pisani and co-workers' could show an association between days of delirium and mortality; - each additional day spent in delirium is associated with a 20% increased risk of prolonged hospitalization - translating to over 10 additional days - and a 10% increased risk of death.The reported prevalence of delirium in critically ill patients ranges widely from 11% to 87%. The aim of our study is to investigate the implementation rate of routine delirium assessment in European ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Patients staying in the ICU on the 25th of January (one-day prevalence study)

No exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients
Sampling Method: Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Implementation rate of routine delirium assessment | 24 hours

SECONDARY OUTCOMES:
Point prevalence of ICU delirium | 24 hours
Methodology of delirium assessment (e.g. type of score, frequency of evaluation) | 24 hours
Non-pharmacological treatment-/prevention strategies | 24 hours
Drugs used for delirium treatment | 24 hours
Sedation practices (e.g. scales, daily sedation goals, SBT - spontaneous breathing trials, SAT - spontaneous awakening trials) | 24 hours
Analgesia regimes (e.g. scales) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Study Director — Charité - Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Luetz A, Balzer F, Radtke FM, Jones C, Citerio G, Walder B, Weiss B, Wernecke KD, Spies C. Delirium, sedation and analgesia in the intensive care unit: a multinational, two-part survey among intensivists. PLoS One. 2014 Nov 14;9(11):e110935. doi: 10.1371/journal.pone.0110935. eCollection 2014. PMID 25398099